CLINICAL TRIAL: NCT01480765
Title: Prospective, Double-blinded, Randomised, Placebo Controlled Trial of Pre-emptive Analgesia to Prevent Pain Following Sternotomy for Cardiac Surgery.
Brief Title: Preventing Pain After Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Reda 007583; 2010-024462-21 (Registry Identifier: EudraCT); 11/H0703/7 (Registry Identifier: UK REC Ref)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Pain; Hyperalgesia; Chronic Illness; Neuropathic Pain
MeSH Terms: conditions — Pain; Hyperalgesia; Chronic Disease; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control: Placebo + Placebo (Placebo Comparator): Placebo capsules and Placebo infusion
  Interventions: Drug: Placebo capsules; Drug: Placebo infusion
- Pregabalin and Placebo infusion (Active Comparator): Pregabalin capsules and Placebo infusion
  Interventions: Drug: Pregabalin; Drug: Placebo infusion
- Pregabalin + Ketamine infusion (Active Comparator): Pregabalin capsules + Ketamine infusion
  Interventions: Drug: Pregabalin; Drug: Ketamine infusion

INTERVENTIONS:
Drug: Pregabalin — 150mg (2hrs) pre operatively and twice daily post operatively for 10 days, followed by dose reduction to 75mg twice daily for 2 days and finally to 50 mg twice daily for 2 days
  Arms: Pregabalin + Ketamine infusion; Pregabalin and Placebo infusion
Drug: Ketamine infusion — 0.1mg/kg/hr for 48 hours post operatively
  Arms: Pregabalin + Ketamine infusion
Drug: Placebo capsules — Single capsule (2hrs) pre operatively and twice daily post operatively for 10 days, followed by dose reduction to single capsule twice daily for 2 days and finally to single capsule twice daily for 2 days
  Arms: Control: Placebo + Placebo
Drug: Placebo infusion — Normal saline placebo intravenous infusion for 48 hours
  Arms: Control: Placebo + Placebo; Pregabalin and Placebo infusion

SUMMARY:
The use of pre-emptive analgesia to prevent pain following sternotomy for cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* First time sternotomy for all cardiac surgery
* Patient aged 18 - 80 years

Exclusion Criteria:

* Emergency surgery (decision to operate taken on the day of surgery)
* Previous sternotomy
* Preoperative renal failure (eGFR <60 ml/min)
* History of chronic non-anginal pain
* Chronic pain medication other than paracetamol and non-steroidal anti-inflammatory drugs
* Concurrent use of oxycodone, lorazepam, or ethanol.
* Concurrent use of any drugs for neuropathic pain e.g. antiepileptics, antidepressants
* Allergy to pregabalin, gabapentin or ketamine
* Pregnancy
* Limited understanding of numerical scoring scales
* Previous participation in other trials investigating analgesic agents or any IMP in previous three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-12-12; Primary Completion 2013-03-07 (Actual); Study Completion 2013-03-07 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) pain score (around sternotomy incision site) post surgery, at rest and following 3 maximal coughs. | 3 and 6 months post sternotomy

SECONDARY OUTCOMES:
Total morphine consumption at 24 hours post surgery | 24 hours post surgery
Visual Analogue Scale (VAS) scores at 24 hrs post surgery, at rest and following 3 maximal coughs | 24 hours post surgery
Sedation (including pCO2) and nausea scores at 24 hours post surgery | 24 hours post surgery
Side effect episodes (dizziness, confusion, blurred vision) | First 48 hours
Time to extubation | Post op recovery period
Length of stay in intensive care and hospital | Post operative - acute
28 day mortality | 28 days post surgery
Neuropathic pain score | 3 and 6 months post surgery
  S-LANSS (Short form Leeds Assessment of Neuropathic Symptoms and Signs)
Quality of Life | 3 and 6 months
  EQ-5D validated scoring scale
Survival | 3 and 6 months
QST measurements | Pre op and post op at 72hrs and 3 months
  Pain Pressure Thresholds (PPT) using algometry, both pre and post Diffuse Noxious Inhibitory Control (DNIC) Tactile and Pain Detection Thresholds with mechanical static stimulus using Von Frey hairs (VFH) Dynamic assessment of temporal summation and secondary hyeralgesia with VFH

CONTACTS AND LOCATIONS:
Overall Officials: Sibtain Anwar, MA MB FRCA, Study Director — Barts and The London NHS Trust
Locations (1):
- Pain and Ananesthesia Research Centre, Barts and The London NHS Trust, London, United Kingdom